CLINICAL TRIAL: NCT03782493
Title: Maximizing Outcomes for Preschoolers With Developmental Language Disorder: Testing the Effects of a Sequentially Targeted Naturalistic Intervention.
Brief Title: Maximizing Outcomes for Preschoolers With Developmental Language Disorders
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Vanderbilt University (Other); University of Illinois at Urbana-Champaign (Other)
Responsible Party: Principal Investigator, Megan Roberts, Jane Steiner Hoffman and Michael Hoffman Assistant Professor of Communication Sciences and Disorders, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: U0046320
Record Dates: First submitted 2018-12-10; First posted 2018-12-20 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Developmental Language Disorder
MeSH Terms: conditions — Language Development Disorders

STUDY DESIGN:
Intervention Model Description: A stratified randomized clinical trial design will be used with site (Vanderbilt, Northwestern) and biological sex (boys, girls) as stratification factors and EMT-SF or business-as-usual (BAU) control as a randomization factor.
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessors and data coders will be blind to experimental condition
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Milieu Teaching-Sentence Focus (Experimental): The study intervention is a behavioral intervention which will include individually teaching caregivers to use the intervention strategies from the Enhanced Milieu Teaching-Sentence Focus (EMT-SF) intervention using a manualized protocol (Teach-Model-Coach-Review). Caregivers will participate in 66 intervention sessions across 18 months, targeting vocabulary and grammar as well as the transition to decontextualized language.
  Interventions: Behavioral: the Enhanced Milieu Teaching-Sentence Focus
- Business-as-usual control (No Intervention): Caregivers in the control group will participate in community-based intervention services and receive the same printed intervention instructions, books, and toys at the same intervals as the treatment group, but will not receive EMT-SF intervention.

INTERVENTIONS:
Behavioral: the Enhanced Milieu Teaching-Sentence Focus — Caregivers in the treatment group (EMT-SF) will receive 66 EMT-SF intervention sessions at home over 18 months. They will be taught the intervention strategies using a manualized protocol (Teach-Model-Coach-Review).
  Other Names: EMT-SF
  Arms: Enhanced Milieu Teaching-Sentence Focus

SUMMARY:
The objective of the proposed study is to evaluate the efficacy of the Enhanced Milieu Teaching-Sentence Focus (EMT-SF) intervention, implemented by caregivers and interventionists, relative to a control condition enrolling 108 30-month-old children and their caregivers. The central hypothesis is that intervention will result in better overall child language skills at 49 months of age.

DETAILED DESCRIPTION:
A multi-site, phase 2, randomized clinical trial will be used to determine whether communication support strategies are effective for improving language outcomes in children with emergent developmental language disorder.

At study entry, 108 children with emergent developmental language disorder (DLD) at 30 months of age will be randomly assigned 1:1 to either the EMT-SF treatment condition or a Business as Usual (BAU) control group. The control group is necessary to determine the efficacy of the EMT-SF intervention. The EMT-SF group is necessary to evaluate the effects of systematically teaching caregivers to use these strategies. Because all children in the study have language delays that will make them eligible to receive the early intervention services through the state early intervention program, children in both experimental conditions will receive state-provided community-based intervention according to their Individualized Family Service Plan - the current standard of care or from private speech language therapy providers. Children in the EMT-SF condition will receive an additional 18 months of interventionist plus caregiver-implemented intervention sessions. Children in both groups will be assessed at the start of the study and every 3 months until the child is 49 months old. The goal is to enroll all children at 30 months of age and provide a minimum of 60 of the planned 66 sessions of intervention to each child in the treatment condition; however, variability in age at study entry (e.g., 30 months), intervention dosage, and number of assessment data points will be addressed in the statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Parent or caregiver (mother, father, grandparent) willing to participate in caregiver training over the full 18 months of the study
* Normal non-verbal cognitive abilities
* Receptive and expressive language delay:
* English as the only language spoken to the child in the home
* Provision of signed and dated informed consent form
* Attempts to imitate 10 words

Exclusion Criteria:

* Diagnosis of a neurodevelopmental disability other than DLD (e.g., Down syndrome, ASD, intellectual disability)
* Caregiver report of a major medical condition (e.g., seizures, cancer, stroke, traumatic head injury, cleft lip/palate, cerebral palsy, legally blind, any genetic diagnosis associated - - Caregiver report of preterm birth (i.e., < 37 weeks gestation)
* Caregiver report of hearing impairment or audiological testing indicating hearing thresholds > 20dB
* Caregiver report or direct observation of any problems chewing, sucking through a straw, or blowing bubbles.

Ages: 27 Months to 31 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 108 (Actual)
Dates: Start 2019-04-04 (Actual); Primary Completion 2025-02-22 (Actual); Study Completion 2025-02-22 (Actual)

PRIMARY OUTCOMES:
Clinical Evaluation of Language Fundamentals Preschool - 2nd edition (CELF-P2) | 49 months
  CELF-P2 core language score at 49 months. The core language score includes summing the scaled scores from the following subtests: Word Structure (raw score min = 0; max = 24), Sentence Structure (raw score min = 0; max = 22), and Expressive Vocabulary (raw score mix = 0; max = 40), and deriving a standardized composite score (min = 45; max = 155). These three subtests provide the best diagnostic accuracy between children with and without developmental language disorders. Thus, the Core Language Score is considered the most representative reflection of a child's overall language skills. Higher standard scores represent better language outcomes.
Change in number of different spoken words from a Language Sample | Change between 30 to 49 months (measured every 3 months)
  Slope of total number of different spoken word (NDW) roots from a Language Sample measured every 3 months from 30 to 49 months derived from a 20-minute language sample. Higher scores represent better language outcomes.
Change in a latent factor of grammar from a Language Sample | Change between 30 to 49 months (measured every 3 months)
  Change in a latent variable of number of different verbs, number of different subjects, tense/agreement productivity, index of productive syntax, clauses per utterance derived from a 20-minute language sample. Higher scores represent better language outcomes.

SECONDARY OUTCOMES:
Peabody Picture Vocabulary Test - 5th Edition (PPVT-5) | 36 months
  PPVT standard score (min = 20, max = 160). Higher scores represent better outcomes.
Expressive Vocabulary Test - 3rd edition (EVT-3) | 36 months
  Expressive Vocabulary Test (EVT-3) standard score (min = 20; max = 160). Higher scores represent better outcomes.
Structured Photographic Expressive Language Test - Preschool 2nd edition (SPELT-P2) | 42 months
  Structured Photographic Expressive Language Test (SPELT P-2) raw score (min = 0; max = 40). Higher scores represent better outcomes.
Structured Photographic Expressive Language Test - Preschool 2nd edition (SPELT-P2) | 49 months
  Structured Photographic Expressive Language Test (SPELT P-2) raw score (min = 0; max = 40). Higher scores represent better outcomes.
Test of Early Grammatical Impairment - 3rd person singular & past tense probes (TEGI) | 42 months
  Test of Early Grammatical Impairment (TEGI) raw score for subscales: Third Person Singular Probe subscale (min = 0; max = 10) and the Past Tense Probe subscale (min = 0; max = 18). Higher scores represent better outcomes.
Test of Early Grammatical Impairment - 3rd person singular & past tense probes (TEGI) | 49 months
  Test of Early Grammatical Impairment (TEGI) raw score for subscales: Third Person Singular Probe subscale (min = 0; max = 10) and the Past Tense Probe subscale (min = 0; max = 18). Higher scores represent better outcomes.
Focus on the Outcomes of Children Under Six (FOCUS) | 49 months
  Focus on the Outcomes of Children Under Six (FOCUS) total raw score (min = 0, max = 350). Higher scores represent better outcomes.
Decontextualized language from a Language Sample | 49 months
  Total number of utterances that contain decontextualized language from a 20-minute Language Sample. Higher scores represent better language outcomes.
Renfrew Bus Story - North American Edition (RBS-NA) | 49 months
  Information score (min = 0; max = 52) from the Renfrew Bus Story. Higher scores represent better outcomes.
Child Behavior Checklist (CBCL) | 49 months
  Child Behavior Checklist Internalizing T score (min = 29; max = 100). Lower scores represent better outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Megan Y Roberts, PhD, Principal Investigator — Northwestern University; Pamela Hadley, PhD, Principal Investigator — University of Illinois at Urbana-Champaign; Ann Kaiser, PhD, Principal Investigator — Vanderbilt University
Locations (2):
- United States (2):
  - Northwestern University, Evanston, Illinois
  - Vanderbilt University, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
Transcripts from caregiver-child and examiner-child language samples will also be donated to the Child Language Data Exchange System (http://childes.psy.cmu.edu), an international repository of child language data. Access to the data will be openly available. Researchers who access the transcripts will be expected to abide by the established guidelines for use of TalkBank data http://talkbank.org/share/irb/options.html.
Access Criteria: Data and associated documentation available to users only under a data-sharing agreement that provides for a commitment: (1) to use the data only for research purposes and not to identify any individual participant; (2) to secure the data using appropriate computer technology; (3) to destroy or return the data after analyses are completed; and (4) to cite the grant and key publications describing the database and measures in any resulting presentations and publications.

DOCUMENTS (1):
  • Informed Consent Form (2021-08-19): https://cdn.clinicaltrials.gov/large-docs/93/NCT03782493/ICF_000.pdf